CLINICAL TRIAL: NCT06442098
Title: Camp SMART Speech to Print Summer Literacy Camp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HS-2024-0077
Record Dates: First submitted 2024-05-09; First posted 2024-06-04 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Reading Disorder, Developmental
Keywords: Literacy Intervention
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: Alternating Treatment Single Subject Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Code First (Experimental): Children in this condition will receive 7 sessions of code-focused reading intervention followed by 7 sessions of morphology-focused reading intervention.
  Interventions: Behavioral: CAMP SMART Literacy Summer Camp
- Morphology First (Experimental): Children in this condition will receive 7 sessions of morphology-focused reading intervention followed by 7 sessions of code-focused reading intervention.
  Interventions: Behavioral: CAMP SMART Literacy Summer Camp

INTERVENTIONS:
Behavioral: CAMP SMART Literacy Summer Camp — Multimodal approach to reading intervention

SUMMARY:
This project aims to explore the feasibility and efficacy of a 6-week, intensive summer literacy intervention provided to children in 1st-3rd grades.

DETAILED DESCRIPTION:
1. Purpose/objective:

   To determine the feasibility and preliminary effectiveness of a 6-week literacy summer camp for improving language and literacy outcomes of children with identified language or literacy difficulties.
2. Methods:

   This intervention will be provided by students in the speech and hearing clinic on SDSU's campus. The summer clinical sessions last for 8 weeks. Week 1 will be used for the pre-testing of each participant's baseline language (morphological awareness, phonological awareness, morphosyntax, vocabulary, and narrative language skills) and reading (letter knowledge, nonword reading, reading fluency and reading comprehension). In weeks 2-7, the intervention will take place. This will consist of 3, 3-hour sessions per week. Finally, in week 8, the investigators will conduct post-testing of children's language and reading skills.
3. Subjects:

   The investigators will recruit a maximum of 12 students who are in the summer after Kindergarten, first, or second grade. The investigators will be recruiting students from the local community who either a) have IEPs with eligibility of SLI or SLD-reading or b) have documented parent or teacher concern for reading and/or language skills as determined by parent questionnaire.
4. Planned analyses:

Planned analyses will include analysis of improvement in each of the language and reading skills from pre-test to post-test. The investigators will also include probes of performance of reading skills to allow for single subject analysis. The investigators will develop fidelity rubrics to explore the fidelity of intervention implementation and will analyze how fidelity relates to individual-child-level improvement.

ELIGIBILITY:
Inclusion Criteria:

* Students who are in the summer after Kindergarten, first, or second grade.
* Students from the local community who either a) have IEPs with eligibility of SLI or SLD-reading or b) have documented parent or teacher concern for reading and/or language skills as determined by parent questionnaire.
* Children who fit the above criteria will additionally be determined eligible for the intervention based on language or reading composite skills one or more standard deviations below the mean on the Test of Integrated Language and Literacy Skills (TILLS).
* Children who are rising 4th, 5th, or 6th graders and who have an IEP with eligibility of SLI or SLD-Reading and who demonstrate composite scores one or more standard deviations below the mean on the TILLS may be considered if space remains after recruitment of 1st-3rd graders.

Exclusion Criteria:

* Students who do not either a) have an IEP or b) have documented parent or teacher concern based on parent questionnaire.
* Students who score within the typical range on the TILLS.
* Students who are deaf or blind.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Spelling Probes | Children will spell 10 CVC words at the conclusion of each of their 14 intervention sessions. Their performance will be charted and tracked.
  Experimenter-created lists of CVC words that children will be asked to spell

SECONDARY OUTCOMES:
Test of Integrated Language and Literacy Skills standard score | Administered prior to the initiation of the intervention and upon conclusion of the intervention.
  Standardized measure of language and reading skills that assesses real and non-word reading and spelling as well as oral language skills in English.

CONTACTS AND LOCATIONS:
Locations (1):
- SDSU Speech, Language, and Hearing Clnic, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No